CLINICAL TRIAL: NCT03161509
Title: Effect of Sleeve Gastroctomy on Pharmacokinetics of Paracetamol and Antiepileptic Drugs
Brief Title: Pharmacokinetics of Paracetamol and Antiepileptic Drugs After Sleeve Gastrectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: publication of better study
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Irit HOCHBERG MD, Principle investigator, Attending physician in Institute of Endocrinology, Diabetes and Metabolism, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0563-16-RMB
Record Dates: First submitted 2017-04-27; First posted 2017-05-19 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2017-05

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Acetaminophen; Anticonvulsants; Lamotrigine; Phenytoin; Valproic Acid

STUDY DESIGN:
Intervention Model Description: All participants will undergo blood tests for pharmacokinetic of paracetamol before and 6 months after sleeve gastrectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paracetamol (Experimental): 10 participants will undergo measurement of paracetamol levels before and after sleeve gastrectomy
  Interventions: Drug: Paracetamol
- antiepileptic drug (Experimental): Up to 10 participants in each drug (up to 4 medications, total of up to 40 participants) will undergo measurement of levels of their chronic medication after a dose before and after sleeve gastrectomy
  Interventions: Drug: Antiepileptic (either carbamazepine, lamotrigine, phenytoin or valproic acid)

INTERVENTIONS:
Drug: Paracetamol — single dose of 1 gr paracetamol
  Arms: paracetamol
Drug: Antiepileptic (either carbamazepine, lamotrigine, phenytoin or valproic acid) — Single dose of antiepileptic drug (either carbamazepine, lamotrigine, phenytoin or valproic acid) for which the participant is taking chronically in stable dose
  Other Names: Antiepileptic
  Arms: antiepileptic drug

SUMMARY:
Sleeve gastrectomy may affect drug pharmacokinetics in several potential ways. We will measure pharmakokinetics of paracetamol and antiepileptic drugs before and 6 months after sleeve gastrectomy.

DETAILED DESCRIPTION:
Sleeve gastrectomy may affect drug pharmacokinetics in several potential ways. We will measure pharmakokinetics of paracetamol (in consenting subjects that are undergoing sleeve gastrectomy) and antiepileptic drugs (in consenting subjects that are chronically treated by a stable dose) before and 6 months after sleeve gastrectomy in 10 subjects.

Blood tests will be taken for drug levels before and 4-8 times after the subject takes the drug. A pharmacokinetic curve will be calculated and compared for each subject between prior to surgery and after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. BMI over 30 and eligible for sleeve gastrectomy
2. Mentally capable for consent
3. (for the antiepileptic drug intervention) chronic stable treatment of antiepileptic drug

Exclusion Criteria:

1. Gastrointestinal illness impairing absorption
2. renal failure (glomerular filtration rate<45)
3. liver cirrhosis
4. heart failure (New York Heart Association class III or IV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic curve of paracetamol or antiepileptic drug: AUC | 8 hours
  sequential measurement of paracetamol or antiepileptic drug (carbamazepine, lamotrigine, phenytoin or valproic acid), AUC

CONTACTS AND LOCATIONS:
Overall Officials: Irit Hochberg, MD/PhD, Principal Investigator — Rambam Healthcare Campus
Locations (1):
- Rambam Healthcare Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request